CLINICAL TRIAL: NCT04379804
Title: COMPARISON OF THE INCIDENCE OF RECURRENT LARYNGEAL INJURY FOLLOWING THE DISSECTİON OF THE NERVE BY CRANIO-CAUDAL AND LATERAL APPROACH BY USING INTROPERATIVE NERVE MONITORING
Brief Title: CRANIO-CAUDAL AND LATERAL APPROACH FOR RECURRENT LARYNGEAL NERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yalin Iscan, MD, General Surgery Specialist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CranioCaudal
Record Dates: First submitted 2020-04-18; First posted 2020-05-08 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Laryngeal Nerve Injuries
Keywords: cranio-caudal approach; lateral approach; intraoperative nerve monitoring
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Computer generated random numbers were generated and printed on cards. These cards were placed in sealed, opaque envelopes. On the morning of operation, one envelope was opened before the operation and, depending of the parity of the number, RLN's of the patient were dissected either by cranio-caudal or lateral dissection during the operation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral approach (Active Comparator): Following the ligation of upper pole vessels, the thyroid lobe lobe was pulled anteromedially and the RLN was dissected within the carotid triangle at the level of inferior thyroid artery. The tissue between the carotid artery and the trachea was dissected gently parallel to the direction of the nerve until the nerve is identified visually and,or by hand held stimulation probe. After the identification of RLN, the vessels of inferior thyroid lobe was ligated. The nerve was dissected along its course to the entry point, and then the thyroid lobe was totally dissected from the trachea and the lobectomy was completed. If adverse EMG changes were encountered during lateral approach, traction was released immediately and waited for recovery.
  Interventions: Procedure: Lateral approach
- Cranio-caudal approach (Active Comparator): Following the ligation of upper pole vessels, the upper pole was retracted antero-medially to expose crico-pharyngeal muscle. The RLN nerve was identified at the point of entry both visually and with hand held stimulation probe. The RLN dissection was proceeded craniocaudally by the division of the suspensory ligaments of the berry through the level of inferior thyroid artery. After the identification and visualitzation of the RLN through its whole course, the medial and inferior vessels of the thyroid gland were dissected and ligated. Then, the lobe was dissected from the trachea and lobectomy was completed.
  Interventions: Procedure: Cranio-caudal approach

INTERVENTIONS:
Procedure: Lateral approach — Following the ligation of upper pole vessels, the thyroid lobe was pulled anteromedially and the RLN was dissected within the carotid triangle at the level of inferior thyroid artery (ITA).
  Arms: Lateral approach
Procedure: Cranio-caudal approach — Following the ligation of upper pole vessels, the upper pole was retracted antero-medially to expose crico-pharyngeal muscle. The RLN was identified at the point of entry both visually and with hand held stimulation probe
  Arms: Cranio-caudal approach

SUMMARY:
The recurrent laryngeal nerve (RLN) dissection should be performed cranio-caudally in TOETVA approach.The aim of this study was to compare the cranio-caudal and lateral approach for RLN dissection in regard with the rates of LOS during conventional thyroidectomy using continuous intraoperative nerve monitoring (CIONM).

DETAILED DESCRIPTION:
During the thyroid surgery, the identification of the recurrent laryngeal nerve (RLN) and the dissection through its entry point is still the gold standard in prevention of the nerve injury and to decrease the RLN palsy rate. Intraoperative nerve monitoring (IONM) has also so many benefits to search, identify and dissect the nerve through its course during thyroid surgery and especially the most important benefit of the IONM is to have real time information about the function of the RLN. Most of the endocrine surgeons use the inferolateral approach for RLN identification under the guidance of the IONM in the recent years. However after the definition of the transoral endoscopic thyroidectomy vestibular approach (TOETVA) technique, the approach to the RLN have to be changed to craniocaudal approach in which a way that most of the surgeons are not familiar with. The different approaches of the recurrent laryngeal nerve depend on the indications and on the surgeon's habit. Several approaches exist such as the superior approach ,the lateral approach, and the inferior approach.

ELIGIBILITY:
Inclusion criteria:

* Multinoduler Goitre
* Thyroid papillary cancer
* Solitary thyroid nodule

Exclusion criteria:

* previous thyroid or parathyroid surgery,
* substernal goiter,
* preoperative VCP,
* evidence of lateral lymph node metastasis,
* intentional transection of the RLN due to tumor invasion,
* failure to assess RLN functioning due to equipment issues with the IONM setup,
* presurgical dissection amplitude of <500µV,
* patient's refusal to participate

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Recurrent laryngeal nerve injury | 6 months postoperatively
  Gross anatomical injury or functional injury demonstrated by nerve monitoring

SECONDARY OUTCOMES:
Serum levels of calcium | First day postoperatively
  On the first postoperative day to identify hypocalcemia
Serum levels of parathormone | First day postoperatively
  On the first postoperative day to identify hypoparathyroidism
Recovery of EMG changes | 20 minutes after initial EMG changes
  adverse EMG parameters were defined as amplitude decrease of 50% or more of baseline value and,or latency increase of 10% or more

CONTACTS AND LOCATIONS:
Overall Officials: Yalin İscan, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04379804/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04379804/SAP_001.pdf
  • Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04379804/ICF_002.pdf